CLINICAL TRIAL: NCT00475839
Title: A Randomized Trial Comparing the Monarc Subfascial Hammock Procedure With Tension-free Vaginal Tape Procedure for the Surgical Treatment of Stress Urinary Incontinence
Brief Title: Study Comparing Tension-free Vaginal Tape With the Monarc Procedure for Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Good Samaritan Hospital, Ohio (Other); Greater Baltimore Medical Center (Other); American Medical Systems (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCF 7616
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; sling procedures; tension-free vaginal tape; transobturator
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tension-free Vaginal Tape (Active Comparator)
  Interventions: Device: Tension-free Vaginal Tape
- Monarc Sub-fascial hammock (Active Comparator)
  Interventions: Device: Monarc sub-fascial hammock

INTERVENTIONS:
Device: Tension-free Vaginal Tape
  Arms: Tension-free Vaginal Tape
Device: Monarc sub-fascial hammock
  Arms: Monarc Sub-fascial hammock

SUMMARY:
Urinary incontinence is a major health issue in women. It is estimated to affect 30 - 40% of older women. Stress urinary incontinence, the most common form of this disease, is treated primarily with surgery. A woman's lifetime risk of surgery for SUI is 4%, with nearly 1/3 of surgery being performed for recurrences. Many different surgical procedures have been described for the treatment of SUI and there is no general agreement as to the most effective. This study compares the safety and efficacy of the tension-free vaginal tape procedure to the Monarc subfascial hammock procedure in the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence symptoms
* Urodynamic stress incontinence confirmed with multichannel urodynamic testing
* Age of at least 21 years
* Desires surgical correction of stress urinary incontinence

Exclusion Criteria:

* Post-void residual volume >100cc
* Detrusor overactivity on preoperative multichannel urodynamic testing
* History of previous synthetic, biologic or fascial sub-urethral sling
* Desires future childbearing
* Chronic inguinal or vulvar abscess or history of Hidradenitis Suppurativa
* History of bleeding diathesis or current anti-coagulation therapy
* Inguinal lymphadenopathy or inguinal/vulvar mass
* Current genitourinary fistula or urethral diverticulum
* Reversible cause of incontinence (i.e. drug effect)
* Contraindication to surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2004-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The presence of abnormal bladder function, defined as the sign or symptom of urinary incontinence or urinary retention | 12 months

SECONDARY OUTCOMES:
Complications
Postoperative pain | 2 weeks, 6 weeks
HRQOL | 6 months, 12 months, 18 months, 24 months
Sexual function | 12 months, 24 months
Global improvement in bladder function | 6 months, 12 months, 18 months, 24 months
Development of anterior vaginal prolapse | 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Barber, MD, MHS, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Barber MD, Kleeman S, Karram MM, Paraiso MF, Walters MD, Vasavada S, Ellerkmann M. Transobturator tape compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):611-21. doi: 10.1097/AOG.0b013e318162f22e. PMID 18310363